CLINICAL TRIAL: NCT06649045
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Once Daily in Participants Who Have Obstructive Sleep Apnea and Obesity or Overweight: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Master Protocol for Orforglipron in Participants With Obstructive Sleep Apnea and Obesity or Overweight
Acronym: ATTAIN-OSA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27226; J5P-MC-GZRA (Other: Eli Lilly and Company); J5P-MC-GZ01 (Other: Eli Lilly and Company); J5P-MC-GZ02 (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-17; First posted 2024-10-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: OSA; Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally.
  Study 1 GZ01: Participants who are unable or unwilling to use PAP
  Study 2 GZ02: Participants who plan to continue PAP therapy
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants will receive placebo orally.
  Study 1 GZ01: Participants who are unable or unwilling to use PAP
  Study 2 GZ02: Participants who plan to continue PAP therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally.
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
Study GZRA is a master protocol that will support 2 independent studies, GZ01 and GZ02. Participants will be assigned to the appropriate study prior to randomization. The purpose of the studies is to evaluate the efficacy and safety of orforglipron in participants who have moderate-to-severe OSA and obesity or overweight. Study GZ01 will include participants who are unable or are unwilling to use PAP therapy. Study GZ02 will include participants who are on PAP therapy for at least 3 months at time of screening and plan to continue PAP therapy during the study.

ELIGIBILITY:
Inclusion Criteria:

Master GZRA inclusion criteria

* have AHI ≥15 on PSG as part of the trial at screening (V1).
* have body mass index (BMI) ≥27 kg/m²

Study 1 GZ01 inclusion criteria

* Participants who are unable or unwilling to use PAP therapy.
* Participants must not have used PAP for at least 4 weeks prior to screening.

Study 2 GZ02 inclusion criteria

* Participants who have been on PAP therapy for at least 3 consecutive months prior to study start and plan to continue PAP therapy during the study.

Exclusion Criteria:

Master GZRA exclusion criteria

* Have Type 1 diabetes (T1D) or Type 2 diabetes (T2D), history of ketoacidosis, or hyperosmolar state/coma
* Have HbA1c ≥6.5% (≥ 48 mmol/mol), as determined by the central laboratory at Visit 1.
* Had any previous or planned upper airway surgery for sleep apnea or major ear, nose or throat surgery
* Have diagnosis of Central or Mixed Sleep Apnea with % of mixed or central apneas/hypopneas ≥50%, or diagnosis of Cheyne Stokes Respiration
* Diagnosis of Obesity Hypoventilation Syndrome or daytime hypercapnia.
* Active device treatment of OSA other than PAP therapy
* Respiratory and neuromuscular diseases that could interfere with the results of the trial in the opinion of the investigator.
* Have a self-reported change in body weight >5 kg within 3 months prior to screening
* Have a prior or planned surgical treatment for obesity (excluding liposuction, abdominoplasty or cryolipolysis if performed more than 1 year prior to screening)
* Have a prior or planned endoscopic and/or present device-based therapy for obesity.
* Have obesity induced by other endocrinologic disorders or diagnosed monogenetic or syndromic forms of obesity.

Study 2 GZ02 exclusion criteria

* Have personal or job-related responsibilities, or in the opinion of the investigator have any situation that would make it unsafe to stop PAP therapy for 7 days prior to PSG testing during the study.
* Are unwilling to temporary discontinue PAP therapy for 7 days prior to PSG testing during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Apnea-Hypopnea Index (AHI) | Baseline to Week 52

SECONDARY OUTCOMES:
Percent Change from Baseline in AHI | Baseline to Week 52
Change from Baseline in Sleep Apnea-Specific Hypoxic Burden (SASHB) (% min/hour) | Baseline to Week 52
Change from Baseline in Patient-Reported Outcome Measurement Information System (PROMIS) Short Form Sleep-Related Impairment 8a T-score | Baseline to Week 52
Percentage of Participants Achieving ≥50% AHI Reduction | Baseline to Week 52
Percent of Participants with AHI<5 or with AHI 5-14 with Epworth Sleepiness Scale (ESS) ≤10 | Baseline to Week 52
Percent Change from Baseline in Body Weight | Baseline to Week 52
Change from Baseline in high-sensitivity C reactive protein (hsCRP) Concentration | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (66):
- United States (15):
  - Ark Clinical Research, Long Beach, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Care Access - Aurora, Aurora, Colorado
  - EBGS Clinical Research Center, Snellville, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Care Access - Shreveport, Shreveport, Louisiana
  - The Sleep Spot - Maimonides, Albuquerque, New Mexico
  - Accellacare - Wilmington, Wilmington, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Prime Revival Research Institute, LLC, Flower Mound, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Argentina (8):
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Centro Privado de Medicina Respiratoria, Paraná
  - Instituto Médico Río Cuarto, Río Cuarto
  - INECO Neurociencias Oroño, Rosario
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
- Brazil (5):
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - CPQuali Pesquisa Clínica, São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Hospital das Clinicas FMUSP, São Paulo
- China (11):
  - Peking University People's Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan Provincial People's Hospital, Chengdu
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Huzhou Central Hospital, Huzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Jiangxi Provincial People's Hospital, Nanchang
  - Ningbo First Hospital, Ningbo
  - Pudong New Area People's Hospital Shanghai, Shanghai
  - ShenZhen People's Hospital, Shenzhen
  - Wuxi People's Hospital, Wuxi
- Czechia (3):
  - Nemocnice Rudolfa a Stefanie Benešov, Benešov
  - Milan Kvapil s.r.o., Diabetologicka ambulance, Prague
  - Praglandia s.r.o, Prague
- Germany (8):
  - CIMS Studienzentrum Bamberg, Bamberg
  - Advanced Sleep Research, Berlin
  - InnoDiab Forschung Gmbh, Essen
  - Unterfrintroper Hausarztzentrum Klinische Forschung, Essen
  - Siteworks GmbH - Hannover, Hanover
  - Siteworks - Karlsruhe, Karlsruhe
  - Institut für Diabetesforschung GmbH Münster, Münster
  - RED-Institut GmbH, Oldenburg
- Japan (5):
  - Kirigaokatsuda Hospital, Kitakyushu
  - Osaka Kaisei Hospital, Osaka
  - Sakai City Medical Center, Sakai
  - Nakamura Clinic, Urasoe
  - RESM Respiratory and Sleep Medical Care Clinic, Yokohama
- Mexico (7):
  - Enclifar Ensayos Clínicos Farmacológicos Sc, Chihuahua City
  - Diseno y Planeacion en Investigacion Medica, Guadalajara
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali
  - RM Pharma Specialists - Unidad Especializada en Datos, Mexico City
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City
  - CEINV Salud, Monterrey
- Taiwan (4):
  - Chiayi Christian Hospital, Chiayi City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/